CLINICAL TRIAL: NCT03322241
Title: Medical Provider Experience and Assessment On Healthcare Decisions Post-Testing On Risk Reducing, and Preventative Strategies Utilizing Wellness Lab Tests
Brief Title: Increase Surveillance for Wellness Decisions, Also to Determine Targeted Risk-reducing and Preventative Strategies
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Data Collection Analysis Business Management (Other)
Collaborators: PAS Research Services (Other)
Responsible Party: Sponsor
Other Study IDs: PAS1464
Record Dates: First submitted 2017-10-24; First posted 2017-10-26 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Overall Wellness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: overall wellness — Wellness lab testing

SUMMARY:
Healthcare Decisions Post-Testing On Risk Reducing, and Preventative Strategies Utilizing Wellness Lab Tests

DETAILED DESCRIPTION:
The general design of this study is collecting data and reviewing the Principal Investigators' Standard Operating Procedures on wellness testing and changes made to their specific SOP.

ELIGIBILITY:
Inclusion Criteria:

* Must be a Medical Practitioner

  * Medical Doctor (MD)
  * Doctor of Osteopathic (DO)
  * Physician Assistant (PA)
  * Advanced Practice Registered Nurse (APRN)
  * Nurse Practitioner (NP)
* Must have a current standard operating procedure that includes obtaining/reviewing medical history and family medical history.

Exclusion Criteria:

* Government-funded insurance data cannot be included in the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Current standard operating procedures for providers
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-05-04 (Actual); Primary Completion 2020-05-04 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Provider Structures and Processes | 36 months
  Plan of Care Changes due to Wellness testing. Provider based observational survey system on the health and well-being of patients and populations

CONTACTS AND LOCATIONS:
Locations (1):
- DCABM, Land O' Lakes, Florida, United States